CLINICAL TRIAL: NCT02468856
Title: Effect of Armodafinil on Simulated Driving, Electroencephalogram and Cognitive Performance in Sleep Deprived Healthy Subjects
Brief Title: Effect of Armodafinil on Simulated Driving
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: IRB201500170; OCR16236 (Other: University of Florida)
Record Dates: First submitted 2015-05-26; First posted 2015-06-11 (Estimated); Last update posted 2018-12-31 (Actual); Status verified 2018-12

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — Modafinil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Armodafinil (Active Comparator): Armodafinil 250 mg tablets, one time administration per study session in the morning of day 2
  Interventions: Drug: armodafinil
- Placebo (Placebo Comparator): one time administration per study session in the morning of day 2
  Interventions: Drug: Placebo (for armodafinil)

INTERVENTIONS:
Drug: armodafinil — Armodafinil 250 mg tablet single dose administration. Outcome measures: Driving simulator performance, Electroencephalogram activity, Area under the plasma concentration versus time curve (AUC), Motor Praxis Task, the Visual Object Learning Test, the Fractal-2-Back, the Abstract Matching, the Line Orientation Test, the Digit-Symbol Substitution Task, the Balloon Analog Risk Test, and the Psychomotor Vigilance Test
  Other Names: Nuvigil
  Arms: Armodafinil
Drug: Placebo (for armodafinil) — Placebo tablet single dose administration. Outcome measures: Driving simulator performance, Electroencephalogram activity, Motor Praxis Task, the Visual Object Learning Test, the Fractal-2-Back, the Abstract Matching, the Line Orientation Test, the Digit-Symbol Substitution Task, the Balloon Analog Risk Test, and the Psychomotor Vigilance Test
  Arms: Placebo

SUMMARY:
Sleep deprivation slows reaction time, reduces vigilance and impairs judgment and information processing. Chronic effects include metabolic dysfunction, cardiovascular disease and cancer. Sleep deprivation affects quality of life when it causes errors in judgment, whether these occur behind the wheel of an automobile or in a hospital. Armodafinil, a non-amphetamine wakefulness promoting medication, indicated for excessive sleepiness associated with obstructive sleep apnea, narcolepsy, and shift work sleep disorder is used to mitigate the effects of sleep deprivation.

This study will characterize the effect of armodafinil on driving simulator performance. The effects of armodafinil compared to placebo will be studied in a double blind crossover trial involving 10 healthy subjects with serial assessments at baseline and after extensive sleep deprivation. Using simultaneous electroencephalogram (EEG) recording during simulated driving and neurocognitive assessments of vigilance, the relationship between brain activity and cognitive performance will be established.

DETAILED DESCRIPTION:
On the first study day, the subjects will come to the Clinical Research Center (CRC) early in the morning. In the first 90 minutes (acclimation session) of the study day EEG electrodes will be applied and EEG signals will be measured continuously throughout the session. Subjects will be instructed of the controls and operation of the driving simulator and perform a 10 minute test drive to familiarize with it. Afterwards they will perform a battery of cognitive tests including the Motor Praxis Task, the Visual Object Learning Test, the Fractal-2-Back, the Abstract Matching, the Line Orientation Test, the Digit-Symbol Substitution Task, the Balloon Analog Risk Test, and the Psychomotor Vigilance Test to get familiar with the cognitive tests. The cognitive battery will last approximately 25 minutes. The collected data of the conditioning session won't be part of the analysis. The purpose of the session is that subjects adapt to the measures.

Following the acclimation session, the resting baseline for the subjects will be measured which will consist of a simultaneous assessment of cognitive performance and brain activity. The subjects will first drive for 30 minutes on the driving simulator to establish a resting baseline of the driving performance. Afterwards a resting baseline for cognitive tests will be established to measure attention, vigilance, risk-taking and decision-making. EEG will be recorded concurrently during driving and cognitive tests. No blood samples will be taken during the assessment of the resting baseline. Subjects will be discharged from the CRC after completion of the baseline session (approximately 2 hours) until the evening. During this time subjects are not allowed to sleep and they will be informed to not consume any caffeine containing products (e.g. Red Bull, coffee). Upon return to the CRC, the subjects will be sleep deprived and supervised by at least one of the study coordinators and at least one additional person to make sure the subjects don't fall asleep during the night.

The following day, 24 hours after the resting baseline session, the fatigue baseline session will start. Sessions of resting baseline and fatigue baseline will be scheduled for the same time of day on two consecutive days to account for circadian alignment. The testing procedure will be identical to the resting baseline session that means subjects will drive for 60 minutes on the driving simulator and perform the same cognitive tests as in the baseline session. After completion of the fatigue baseline session, the study drug (armodafinil 250 mg or placebo) will be administered. To determine the pharmacokinetics, blood samples will be obtained prior to drug dosing and at 0.5, 1, 1.5, 2, 3, 4, 6, 8 and 10 hours post-dose through an intravenous catheter placed in the arm vein of the subjects. After study drug intake subjects will perform 5 sessions on the driving simulator consisting of 30-minute drives. The same battery of tests performed at baseline will be performed between the drives. The tested cognitive abilities play an important role during driving and the investigators will investigate to what extent sleep deprivation alters these abilities and how armodafinil is able to counter the deteriorating effects of sleep deprivation on these capabilities.

ELIGIBILITY:
Inclusion criteria

1. Male or females, between age 18 and 35 years of age, inclusive.
2. Body mass index (BMI) from 18.5 to 29.9 kg/m2, inclusive.
3. A valid driver's license.
4. Healthy on the basis of physical examination, medical history, vital signs.
5. Absence of clinically significant abnormalities in the subject's sleep history. The study physician will base this decision on the Epworth Sleepiness Scale and a discussion with the subject about his or her sleep history.
6. Female subjects must be postmenopausal (for at least 6 months), surgically sterile, or abstinent; or, if of childbearing potential and sexually active, be practicing an effective method of birth control (e.g., intrauterine device, double-barrier method, male partner sterilization) before entry and throughout the study; have a negative urine pregnancy test at screening, and a negative urine pregnancy test prior to each experimental session. Steroidal contraceptives have been shown to interact with the study drug and are not an acceptable form of contraception for this study (subjects taking steroidal contraceptive drugs are ineligible for this study).
7. Agree not to consume any alcohol 24 hours prior to any study session and until discharge from the unit.
8. Agree not to consume any grapefruit or grapefruit juice 24 hours prior to dosing and until discharge from the unit.
9. Agree not to use armodafinil or modafinil-containing medications 2 weeks prior to or during any study session (aside from what is administered for the study).
10. Agree not to use any other medication that acts on the central nervous system (prescription or nonprescription) 1 week prior to or during any study session (caffeine is the only exception, subjects are recommended to avoid caffeine for one week prior to a study session, but are required to avoid caffeine for 24 hours prior to and during a study session).
11. The subject is able to understand and comply with protocol requirements, instructions and protocol-stated restrictions and is likely to complete the study as planned. Subject is willing to provide informed consent.

Exclusion criteria

1. History of current significant medical illness including (but not limited to) cardiovascular thrombotic events, myocardial infarction, stroke or other cardiac disease, hypertension, peptic ulcer disease or gastrointestinal bleeding, hematological disease, bronchospastic respiratory disease, asthma, diabetes mellitus, renal or hepatic insufficiency, psychiatric disorders, or any other illness that the investigator considers should exclude the subject.
2. Subjects who have a clinically significant sleep abnormality.
3. Subjects who are shift workers.
4. Evidence of use of drugs of abuse (including but not limited to barbiturates, opiates, cocaine, cannabinoids, amphetamines, and benzodiazepines) assessed via questioning the subject.
5. Subjects that are a smoker and smoke more than 10 cigarettes per day.
6. Known allergies or hypersensitivity to armodafinil or modafinil.
7. The subject has contraindications to take armodafinil.
8. Clinically significant abnormal physical examination, vital signs (e.g. systolic blood pressure>140 mmHg, diastolic blood pressure>90 mmHg, heart rate >100 bpm and <45 bpm) or 12-lead ECG (e.g. corrected QT>450 msec) at screening or abnormal vital signs prior to study drug dosing.
9. The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
10. Pregnant or breast-feeding.
11. Taking a steroidal contraceptive drug or drugs.
12. Donation of 1 or more units (approximately 450 mL) of blood or acute loss of an equivalent amount of blood within 60 days prior to study drug administration.
13. Recent history of surgery; within the past 3 months prior to screening.
14. Clinically significant acute illness within 7 days prior to study drug administration.
15. Strenuous exercise that is more excessive than their normal routine, 48 hours prior to each session, until they are discharged from the unit.
16. Any condition that, in the opinion of the investigator, would compromise the well-being of the subject or the study or prevent the subject from meeting or performing study requirements.
17. Unwillingness or inability to follow the procedures outlined in the protocol.
18. Employees of the investigator or study center, with direct involvement in the proposed study or other studies under the direction of that investigator or study center, as well as family members of the employees or the investigator.
19. Subjects living outside of Gainesville

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2017-05-21 (Actual); Primary Completion 2017-11-30 (Actual); Study Completion 2017-11-30 (Actual)

PRIMARY OUTCOMES:
Effect of armodafinil on simulated driving | Change in resting baseline (Day 1) to fatigue baseline (Day 2).
  Driving performance will primarily be assessed by the standard deviation of the lateral position in centimeter measured by the driving simulator software.
Electroencephalogram activity assessment change in hours post-dose | 0, 1, 2, 4, 5, 6, 8, 9 change in hours post-dose
  Brain activity will be assessed by the electroencephalogram spectral power in microvolt
  ^2.
Driving simulator performance assessment change in hours post-dose | 0, 2, 5, 7.5 change in hours post-dose
  Driving performance will primarily be assessed by the standard deviation of the lateral position in centimeter measured by the driving simulator software.
Effect of armodafinil on electroencephalogram activity | Change in resting baseline (Day 1) to fatigue baseline (Day 2).
  Brain activity will be assessed by the electroencephalogram spectral power in microvolt
  ^2.
Area under the plasma concentration versus time curve (AUC) of armodafinil 250 mg | 0, 0.5, 1, 1.5, 2, 3, 4, 6, 7.5 and 10 hours post-dose

SECONDARY OUTCOMES:
Motor Praxis Task assessment pre-dose | Change in resting baseline (Day 1) to fatigue baseline (Day 2).
  Efficiency Score calculated by the Cognition Software
Motor Praxis Task assessment change in hours post-dose | 1, 4, 6, 9 change in hours post-dose
  Efficiency Score calculated by the Cognition Software
Visual Object Learning Test assessment pre-dose | Change in resting baseline (Day 1) to fatigue baseline (Day 2).
  Efficiency Score calculated by the Cognition Software
Visual Object Learning Test assessment change in hours post-dose | 1, 4, 6, 9 change in hours post-dose
  Efficiency Score calculated by the Cognition Software
Fractal-2-Back assessment pre-dose | Change in resting baseline (Day 1) to fatigue baseline (Day 2).
  Efficiency Score calculated by the Cognition Software
Fractal-2-Back assessment change in hours post-dose | 1, 4, 6, 9 change in hours post-dose
  Efficiency Score calculated by the Cognition Software
Abstract Matching assessment pre-dose | Change in resting baseline (Day 1) to fatigue baseline (Day 2).
  Efficiency Score calculated by the Cognition Software
Abstract Matching assessment change in hours post-dose | 1, 4, 6, 9 change in hours post-dose
  Efficiency Score calculated by the Cognition Software
Line Orientation Test assessment pre-dose | Change in resting baseline (Day 1) to fatigue baseline (Day 2).
  Efficiency Score calculated by the Cognition Software
Line Orientation Test assessment change in hours post-dose | 1, 4, 6, 9 change in hours post-dose
  Efficiency Score calculated by the Cognition Software
Digit-Symbol Substitution Task assessment pre-dose | Change in resting baseline (Day 1) to fatigue baseline (Day 2).
  Efficiency Score calculated by the Cognition Software
Digit-Symbol Substitution Task assessment change in hours post-dose | 1, 4, 6, 9 change in hours post-dose
  Efficiency Score calculated by the Cognition Software
Balloon Analog Risk Test assessment pre-dose | Change in resting baseline (Day 1) to fatigue baseline (Day 2).
  Efficiency Score calculated by the Cognition Software
Balloon Analog Risk Test assessment change in hours post-dose | 1, 4, 6, 9 change in hours post-dose
  Efficiency Score calculated by the Cognition Software
Psychomotor Vigilance Test assessment pre-dose | Change in resting baseline (Day 1) to fatigue baseline (Day 2).
  Efficiency Score calculated by the Cognition Software
Psychomotor Vigilance Test assessment change in hours post-dose | 1, 4, 6, 9 change in hours post-dose
  Efficiency Score calculated by the Cognition Software

CONTACTS AND LOCATIONS:
Overall Officials: Hartmut Derendorf, PhD, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Clinical and Translational Science Institute, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided